CLINICAL TRIAL: NCT05358535
Title: Propofol and Etomidate Admixtures Comparisons Trial (PEAC Trial)
Acronym: PEAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Choi, Assistant Professor of Anesthesiology and Pain Management, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2022-0377
Record Dates: First submitted 2022-04-21; First posted 2022-05-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Propofol Adverse Reaction; Etomidate Adverse Reaction; Anesthesia Complication; Anesthesia; Adverse Effect; Anesthesia; Reaction
Keywords: anesthesia; anesthesiology; adverse drug reaction; drug side effect; sedation; cardiopulmonary; hemodynamics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Propofol; Etomidate

STUDY DESIGN:
Intervention Model Description: This a prospective double blind randomized controlled clinical trial. The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital endoscopy lab.
Who Masked: Participant, Care Provider
Masking Description: Blinding plan: Either the investigational drug service with the CUH central pharmacy will prepare the admixture syringes or a separate anesthesia staff not involved in subject's case will prepare admixture syringes thus preventing any case personnel involved with subject's case or subject from knowing which admixture is present within syringes for subject's case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2) (Experimental): This a prospective double blind randomized controlled clinical trial. The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital endoscopy lab.
  Interventions: Drug: Admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2)
- Admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7) (Experimental): This a prospective double blind randomized controlled clinical trial. The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital endoscopy lab.
  Interventions: Drug: Admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7)

INTERVENTIONS:
Drug: Admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2) — The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital (CUH) endoscopy lab (Endo).
  The objectives are to compare the treatment arms, P2E7 and P7E2, in a randomized controlled double-blind trial for anesthesia for endoscopic procedures. Comparison between an admixture of Propofol/Etomidate 75%/25% versus 25%/75% being utilized as principal anesthetic for endoscopic procedures at CUH endoscopy lab.
  Other Names: propofol; etomidate; P7E2; propofol 75% by volume; etomidate 25% by volume
  Arms: Admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2)
Drug: Admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7) — The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital (CUH) endoscopy lab (Endo).
  The objectives are to compare the treatment arms, P2E7 and P7E2, in a randomized controlled double-blind trial for anesthesia for endoscopic procedures. Comparison between an admixture of Propofol/Etomidate 75%/25% versus 25%/75% being utilized as principal anesthetic for endoscopic procedures at CUH endoscopy lab.
  Other Names: propofol; etomidate; P2E7; propofol 25% by volume; etomidate 75% by volume
  Arms: Admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7)

SUMMARY:
The purpose of this study is to evaluate the hemodynamics and adverse event profile in comparison between two treatment arms, one using an admixture of propofol and etomidate at a ratio by volume of 25%/75% (P2E7), and one using an admixture of propofol and etomidate at a ratio by volume of 75%/25% (P7E2), for anesthesia during endoscopic procedures at the Clements University Hospital (CUH) endoscopy lab (Endo).

DETAILED DESCRIPTION:
Procedural/Surgical anesthesia induction, administration and maintenance with propofol combined with etomidate is commonly used in routine clinical practice in patient with compromised cardiopulmonary status. However, there is no definitive trend or understanding from the literature to discern which ratio of admixture is appropriate for providing stable hemodynamics and minimizing side effects for procedural sedation in gastrointestinal endoscopy procedures. Given the increasing volume for gastrointestinal endoscopy, the increasingly older and greater chronic disease burden of the endoscopic patient population, and the increased utilization of anesthesia for endoscopic procedures this clinical trial aims to provide timely, meaningful and impactful guidance and information for the safe conductance of anesthesia in this patient population.

The objectives are to compare the treatment arms, P2E7 and P7E2, in a randomized controlled double-blind trial for anesthesia for endoscopic procedures. Comparison between an admixture of Propofol/Etomidate 75%/25% versus 25%/75% being utilized as principal anesthetic for endoscopic procedures at CUH endoscopy lab.

Propofol and etomidate can be mixed together in a syringe or similar container for up to 24 hours without adversely affecting appearance, pH, particle size and distribution, zeta potential, observation under centrifugation and drug content and impurity demonstrating the mixture to be physically and chemically compatible. Propofol and Etomidate are both FDA approved for induction and maintenance of general anesthesia in adult patients. Propofol and Etomidate in a wide ranging ratio of combinations in admixture have been utilized for general anesthesia induction and maintenance both in regular standard of care daily clinical practice and within a profound number of research trials including up to a ratio of 80% etomidate and 20 % propofol by volume. Therefore the clinical practice of etomidate and propofol in admixture for the induction and maintenance of general anesthesia in adult patients is standard of care and well founded in the anesthesiology literature. However, there are several important questions about which potential ratio of both drugs provides the best combination of favorable cardiopulmonary effects while having an acceptably low incidence of adverse effects. Thus, this current proposed trial is intended to answer several important questions on that matter.

This trial also will have actual blinding of both patients and practitioners at time of drug administration. Propofol is a white liquid and etomidate is a clear liquid. Thus, past trials where either pure drug was given in sequence or at the same time by separate syringes could not have had any blinding because of this obvious physical quality of the medications. Therefore, only a trial involving an admixture of varying ratios of both drugs could possibly hope to achieve actual blinding as is required for rigorous analysis of results without introducing the bias that comes from a lack of true blinding of patients and practitioners.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years old)
2. Having endoscopic procedure at CUH with anesthesia
3. ASA 3 or above
4. Ejection Fraction test result available

Exclusion Criteria:

1. Known allergies or adverse reactions to study drugs or study drug components or preservatives
2. Patient refusal
3. Clinician refusal
4. Documented cognitive impairments precluding subject ability to consent for themselves unless a surrogate documented legally acceptable decision maker consents for patient participation
5. Prisoner or incarcerated or patients held by law enforcement officials in custody
6. Pregnancy or patient refusal for pregnancy testing or screening (standard UTSW policy and protocol requires pregnancy testing for appropriate patients prior to anesthesia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Time weighted average mean arterial pressure within treatment arm | Throughout entire study estimated to take 6 to 12 months to complete
  Time weighted average mean arterial pressure (every 15 minutes calculate average mean arterial pressure for that interval, then end of case calculate mean of all those means for the entire case)
Average within treatment arm vasopressor use by number of units | Throughout entire study estimated to take 6 to 12 months to complete
  Vasopressor use by number of units (1 unit of vasopressor being defined as 1 unit vasopressor = 100 mcg phenylephrine = 5 mg ephedrine = 0.5 units vasopressin = 5 mcg norepinephrine)4-9 throughout entire intraoperative period (subjects on vasopressor infusions on arrival for endoscopy will not have those vasopressor units added in UNLESS during case, anesthesia clinicians adjust the infusion based on intraoperative clinical situation as well as all bolus doses and new infusions being added as with all other subjects)
Average within treatment arm total minutes under 92% oxygen saturation | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm total minutes under 92% oxygen saturation by pulse oximetry during entire case
% of cases with any MAP below 50 | Throughout entire study estimated to take 6 to 12 months to complete
  % of cases with any MAP below 50
% of cases with any MAP >60% below patient's immediate preoperative MAP | Throughout entire study estimated to take 6 to 12 months to complete
  % of cases with any MAP >60% below patient's immediate preoperative MAP
% of cases with any treatment for Post Operative Nausea and Vomiting | Throughout entire study estimated to take 6 to 12 months to complete
  % of cases with any treatment for Post Operative Nausea and Vomiting
% of cases with any oxygen saturation event below 85% by pulse oximetry | Throughout entire study estimated to take 6 to 12 months to complete
  % of cases with any oxygen saturation event below 85% by pulse oximetry
% of cases with any rapid response or code blue event within 24 hours from anesthesia start | Throughout entire study estimated to take 6 to 12 months to complete
  % of cases with any rapid response or code blue event within 24 hours from anesthesia start
Within treatment arm % of total group with a composite MACE event in the 30 days | Throughout entire study estimated to take 6 to 12 months to complete
  Within treatment arm % of total group with a composite MACE event in the 30 days after starting on day of drug administration
Within treatment arm % of total group with a classic MACE event in the 30 days | Throughout entire study estimated to take 6 to 12 months to complete
  Within treatment arm % of total group with a classic MACE event in the 30 days after starting on day of drug administration
Average within treatment arm antiemetic use by number of doses | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm antiemetic use by number of doses irrespective of antiemetic drug choice
Average within treatment arm time in minutes after dressing complete to discharge | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm time in minutes after dressing complete to discharge to next phase of care or to home from immediate recovery phase of care

SECONDARY OUTCOMES:
Within each treatment arm, average of anesthesia clinicians' assessment of quality | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, average of anesthesia clinicians' assessment of quality of anesthesia during case: Poor, Below Average, Average, Above Average, Excellent (0,1,2,3,4) from all anesthesia staff then average for each treatment arm
Within each treatment arm, average of endoscopists' assessment of quality | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, average of endoscopists' assessment of quality of anesthesia during case: Poor, Below Average, Average, Above Average, Excellent (0,1,2,3,4) from all endoscopy staff then average for each treatment arm
Within each treatment arm, average of patients' assessment of quality | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, average of patients' assessment of quality of anesthesia during case: Poor, Below Average, Average, Above Average, Excellent (0,1,2,3,4) from all patients then average for each treatment arm
Within each treatment arm, number of events of any use of 2 or more | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any use of 2 or more different (beyond study admixtures) sedative or anesthetic adjunct medications
Within each treatment arm, number of events of any use of two or more | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any use of two or more types of antiemetic drugs
Average time in immediate recovery area before discharge to next phase of care | Throughout entire study estimated to take 6 to 12 months to complete
  Average time in immediate recovery area before discharge to next phase of care or to home
Average time from dressing complete to modified Aldrete score >8 | Throughout entire study estimated to take 6 to 12 months to complete
  Average time from dressing complete to modified Aldrete score >8
Within each treatment arm number of composite MACE events in the 30 days | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm number of composite MACE events in the 30 days after starting on day of drug administration
Within each treatment arm number of classic MACE events in the 30 days | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm number of classic MACE events in the 30 days after starting on day of drug administration
Average within treatment arm total dose (mL) of admixture administered | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm total dose (mL) of admixture administered during entire case divided by average time from induction to dressing complete (minutes)
Average within treatment arm total dose (mg) of etomidate during entire case | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm total dose (mg) of etomidate during entire case divided by average time from induction to dressing complete (minutes)
Average within treatment arm total dose (mg) of propofol during entire case | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm total dose (mg) of propofol during entire case divided by average time from induction to dressing complete (minutes)
Average within treatment arm total dose of adjunct sedatives | Throughout entire study estimated to take 6 to 12 months to complete
  Average within treatment arm total dose of fentanyl, sufentanil, midazolam, diphenhydramine, ketamine, morphine, hydromorphone, dexmedetomidine, undiluted propofol, undiluted etomidate (either in mcg or mg as appropriate for each drug) divided by average time from induction to dressing complete (minutes)
Within each treatment arm, number of events of any episode of vomiting | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any episode of vomiting
Within each treatment arm, number of events of any complaint of nausea | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any complaint of nausea
Within each treatment arm, number of events of any syncopal event | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any syncopal event
Within each treatment arm, number of events of any use of one type of antiemetic drug | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any use of one type of antiemetic drug
Within each treatment arm, number of events of any unanticipated admission | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any unanticipated admission, or transfer to higher level of care in the 24 hours after starting on day of drug administration
Within each treatment arm, number of events of any airway adjunct usage | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any airway adjunct usage (oral airway, nasal airway, need for intermittent mask ventilation)
Within each treatment arm, number of events of any use of any additional sedatives | Throughout entire study estimated to take 6 to 12 months to complete
  Within each treatment arm, number of events of any use of any additional sedative or anesthetic adjunct medication (beyond study admixtures) during case (fentanyl, sufentanil, midazolam, diphenhydramine, ketamine, morphine, hydromorphone, dexmedetomidine, undiluted propofol, undiluted etomidate)

CONTACTS AND LOCATIONS:
Overall Officials: Kapil Anand, Study Director — University of Texas
Locations (1):
- Clements University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
1. PHI (name, date of birth, Medical Record number, phone number, email account, admission date)
  2. Demographics (Age, height, weight, BMI)
  3. Medical history
  4. Medication list Intraoperative data collection
     * Time weighted average mean arterial pressure (every 15 minutes calculate average mean arterial pressure for that interval, then end of case calculate mean of all those means for the entire case) Area Under the Threshold for mean arterial pressure (both predefined threshold of 65 mm Hg and for 40% below patient's immediate preoperative MAP)
     * Vasopressor use by number of units (1 unit of vasopressor being defined as 1 unit vasopressor = 100 mcg phenylephrine = 5 mg ephedrine = 0.5 units vasopressin = 5 mcg norepinephrine)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At conclusion of all data analysis and available permanently
Access Criteria: Only study personnel

REFERENCES:
- [Background] Chen L, Liang X, Tan X, Wen H, Jiang J, Li Y. Safety and efficacy of combined use of propofol and etomidate for sedation during gastroscopy: Systematic review and meta-analysis. Medicine (Baltimore). 2019 May;98(20):e15712. doi: 10.1097/MD.0000000000015712. PMID 31096522
- [Background] Yoon SW, Choi GJ, Lee OH, Yoon IJ, Kang H, Baek CW, Jung YH, Woo YC. Comparison of propofol monotherapy and propofol combination therapy for sedation during gastrointestinal endoscopy: A systematic review and meta-analysis. Dig Endosc. 2018 Sep;30(5):580-591. doi: 10.1111/den.13050. Epub 2018 Apr 17. PMID 29526045
- [Background] Hao L, Hu X, Zhu B, Li W, Huang X, Kang F. Clinical observation of the combined use of propofol and etomidate in painless gastroscopy. Medicine (Baltimore). 2020 Nov 6;99(45):e23061. doi: 10.1097/MD.0000000000023061. PMID 33157963
- [Background] Goradia S, Sardaneh AA, Narayan SW, Penm J, Patanwala AE. Vasopressor dose equivalence: A scoping review and suggested formula. J Crit Care. 2021 Feb;61:233-240. doi: 10.1016/j.jcrc.2020.11.002. Epub 2020 Nov 14. PMID 33220576
- [Background] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Background] French WB, Rothstein WB, Scott MJ. Time to Use Peripheral Norepinephrine in the Operating Room. Anesth Analg. 2021 Jul 1;133(1):284-288. doi: 10.1213/ANE.0000000000005558. No abstract available. PMID 33886514
- [Background] Mohta M, Dubey M, Malhotra RK, Tyagi A. Comparison of the potency of phenylephrine and norepinephrine bolus doses used to treat post-spinal hypotension during elective caesarean section. Int J Obstet Anesth. 2019 May;38:25-31. doi: 10.1016/j.ijoa.2018.12.002. Epub 2018 Dec 13. PMID 30685301